CLINICAL TRIAL: NCT06696547
Title: The Effect of Cerebellar Intermittent Theta Burst Stimulation Combined With Conventional Rehabilitation Methods on Gait, Balance, and Disease Anxiety in Patients With Ischemic Stroke
Brief Title: The Effects of Cerebellar Intermittent Theta Burst Stimulation on Gait, Balance, and Disease Anxiety In Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Miray Karamehmetoğlu, M.D., Principal Investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AnkaraCHBilkent-PMR-MK-01
Record Dates: First submitted 2024-11-15; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Hemiplegia Following Ischemic Stroke
Keywords: Stroke; Transcranial Magnetic Stimulation; Gait; Balance
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active CRB-iTBS (Active Comparator): Patients received a total of 30 sessions active CRB-iTBS targeting contralesional lateral cerebellum, 5 days a week for 3 weeks. The cerebellar region to be targeted, on the opposite side of the cerebral lesion, was determined by measuring 3 cm lateral and 1 cm inferior of the inion, which is the anatomical prominence on the occipital bone (3L1I). Stimulation intensity was set at 80% of the active motor threshold (AMT). AMT was defined as the lowest intensity required for a motor-evoked potentials (MEP) above 200 µV in at least 50% of 10 trials when the patient was contracting targeted muscle 10% on the maximum voluntary contraction. Stimulation was administered as 3-burst pulses at a frequency of 50 Hz, with 2-second stimulation repeated every 10 seconds period. This continued for a total duration of 190 seconds, delivering 600 pulses. Each CRB-iTBS session was performed in 2 sessions before daily rehabilitation programs. Thus, 1200 pulses were applied per day.
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham CRB-iTBS (Sham Comparator): Patients received a total of 30 sessions sham CRB-iTBS targeting contralesional lateral cerebellum, 5 days a week for 3 weeks. The cerebellar region to be targeted, on the opposite side of the cerebral lesion, was determined by measuring 3 cm lateral and 1 cm inferior of the inion, which is the anatomical prominence on the occipital bone (3L1I). However, sham coil was used for stimulation. Therefore, no real stimulation was applied to the patients. Instead, a sensation mimicking real stimulation was created through the sham coil, with sounds and sensations on the scalp as if stimulation were occurring. Each sham CRB-iTBS session was performed in 2 sessions before daily rehabilitation programs.
  Interventions: Device: Transcranial Magnetic Stimulation Sham

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Magstim Rapid2 Magnetic Stimulator (Magstim, Whitland Dyfed, UK), 70 mm Figure-of-eight Coil
  Arms: Active CRB-iTBS
Device: Transcranial Magnetic Stimulation Sham — Magstim Rapid2 Magnetic Stimulator (Magstim, Whitland Dyfed, UK), 70 mm Figure-of-eight Sham Coil
  Arms: Sham CRB-iTBS

SUMMARY:
Our study was designed to investigate the effect of cerebellar intermittent theta burst stimulation (iTBS) combined with conventional rehabilitation methods on balance, gait and disease anxiety in patients with ischemic stroke who have residual balance and gait disturbance, using clinical measurement parameters.

DETAILED DESCRIPTION:
Loss of balance and gait functions, which are neurological impairments related to stroke, are among the common functional losses depending on the affected brain region. Reduced independence in daily living activities can lead to increased anxiety during ambulation, risk of falling and fear of falling. Studies have shown that applying theta burst stimulation (TBS) to the cerebellum has long-term effects on the excitability of the cerebello-thalamo-cortical pathways and stimulates synaptic plasticity through various mechanisms. In the literature, there are studies examining the effects of cerebellar iTBS on balance and walking functions in stroke patients, but the number of studies are quite limited.

This study was planned as a prospective, randomized, sham-controlled clinical study. According to the statistical analysis 30 patients who were registered at Ankara Bilkent City Hospital Physical Therapy and Rehabilitation Hospital between February 2022 and April 2023 and met the study criteria were included. The patients were divided into two groups: active (n=15) and sham (n=15). Each group received 30 sessions of either active or sham cerebellar iTBS (CRB-iTBS). Additionally, patients received therapeutic interventions from a physiotherapist, including range of motion exercises, stretching, neurophysiological exercises, balance-coordination training, active-assistive mobilization, and exercises for daily living.

The CRB-iTBS treatment targeted the cerebellum on the opposite side to the cerebral lesions, administered in a total of 30 sessions, twice a day with a 5-minute interval between sessions, over a period of 3 weeks. Each stimulation session consisted of 3-burst pulses at a frequency of 50 Hz, with a 10-second repetitive cycle of 2-second stimulations lasting a total of 190 seconds, delivering 600 pulses per session. Each day, a total of 1200 pulses were administered over two sessions, spaced 5 minutes apart. Patients in the sham CRB-iTBS group received the same protocol with a sham coil that visually resembled the active coil.

Clinical evaluations were conducted three times for each patient: Baseline (before treatment), 3rd week (at the and of treatment), and 6th week.

ELIGIBILITY:
Inclusion Criteria:

* First ischemic stroke,
* Duration between 2 months to 2 years post-stroke,
* Hemiparesis and residual gait and balance disorders related to the lesion in the MCA area (Berg Balance Scale score < 40),
* Lower extremity Brunnstrom value of at least 3 ,
* Mini Mental State Examination ≥ 24,
* Between 18-80 years old

Exclusion Criteria:

* History of seizures,
* Severe general impairmet or concomittant disease,
* Using benzodiazepines, baclofen or antidepressants,
* Having a cardiac pacemaker, cochlear implant, metallic implants in the brain or skull,
* Pregnancy,
* Under 18 or over 80 years old

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) | Baseline (before treatment), 3rd week (at the end of treatment), 6th week
  This is a scale used to evaluate patients' balance during 14 different activities. These activities include: sitting to standig, standing unsupported, sitting unsupported, standing to sitting, transfers, standing unsupported with eyes closed, standing with feet together, reaching forward while standing, picking up an object from the floor, looking back over the shoulder on both the right and left sides, turning 360 degrees, placing a foot on a stool, standing in a toe-heel position, and standing on one foot. The total score after performing the test determines the predicted risk of falls. The minimum score on the test is 0, and the maximum score is 56. Scores are classified as follows: 0-20 indicates a high risk of falling, 21-40 indicates a moderate risk of falling, and 41-56 indicates a low risk of falling.
Gait Analysis- Step Length | Baseline (before treatment), 3rd week (at the end of treatment), 6th week
  The Zebris FDM Type 3 (Zebris Medical GmbH, Germany) device was used to record spatiotemporal data during walking. This system consists of a 3-meter straight platform, with two 1-meter maneuvering platforms at the start and end. It is equipped with sensors and computer software for data analysis. The data collected in the study included step length (cm).
Gait Analysis- Step Width | Baseline (before treatment), 3rd week (at the end of treatment), 6th week
  The Zebris FDM Type 3 (Zebris Medical GmbH, Germany) device was used to record spatiotemporal data during walking. This system consists of a 3-meter straight platform, with two 1-meter maneuvering platforms at the start and end. It is equipped with sensors and computer software for data analysis. The data collected in the study included step width (cm).
Gait Analysis- Walking Speed | Baseline (before treatment), 3rd week (at the end of treatment), 6th week
  The Zebris FDM Type 3 (Zebris Medical GmbH, Germany) device was used to record spatiotemporal data during walking. This system consists of a 3-meter straight platform, with two 1-meter maneuvering platforms at the start and end. It is equipped with sensors and computer software for data analysis. The data collected in the study included walking speed (km/h).

SECONDARY OUTCOMES:
International Falls Efficacy Scale (FES-I) | Baseline (before treatment), 3rd week (at the end of treatment), 6th week
  Patients are evaluated for their level of concern about the risk of falling during 16 different activities. A score of 1 reflects no concern, while a score of 4 reflects a high level of concern. Total scores range from 16 to 64, with higher scores indicating greater anxiety about falling and lower self-confidence during activities.
Barthel Index for Activities of Daily Living (BI) | Baseline (before treatment), 3rd week (at the end of treatment), 6th week
  The Barthel Index (BI) was used to assess physical independence in daily activities on ten-item scale. These items are: feeding, bathing, grooming, dressing, bowels, bladder, toilet use, transfer (bed to chair and back), mobility (on level surfaces). Score of 0 indicating complete dependence and a score of 100 indicating complete independence.
Stroke Specific Quality of Life Scale (SS-QOL) | Baseline (before treatment), 3rd week (at the end of treatment), 6th week
  The Stroke-Specific Quality of Life Scale (SS-QOL) assesses the functionality and quality of life in stroke patients through 49 questions across 12 categories. These categories include: thinking, upper extremity functions, vision, work/productivity, social roles, self-care, personality, mood, mobility, language, family roles, and energy. Scoring is done on a scale from 1 to 5, with a total score ranging from 49 to 245. A score of 49 indicates very low quality of life, while a score of 245 indicates high quality of life.
Hospital Anxiety and Depression Scale (HADS) | Baseline (before treatment), 3rd week (at the end of treatment), 6th week
  Hospital Anxiety and Depression Scale (HADS) consists of 14 questions, which are to be answered based on the patient's experience over the past few days while hospitalized. Seven of the questions assess depression, and seven assess anxiety levels. Separate scoring is done for anxiety and depression. The score may range between 0 and 21 per subscale. Higher scores indicate higher levels of anxiety and depression.

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Acar Sivas, Prof, MD, Study Chair — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No